CLINICAL TRIAL: NCT06536075
Title: Functional Analysis and Antigen Presentation in Striated Ductal Cells of Salivary Glands and Correlation With Sialoscintigraphy in Patients and Animal Models of Sjogren's Syndrome
Brief Title: Functional Analysis of Salivary Glands and Correlation With Sialoscintigraphy in Sjogren's Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Clinical Trial Center, Principal Investigator and visiting staff, National Taiwan University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 202307135MINB
Record Dates: First submitted 2024-07-31; First posted 2024-08-02 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-07

CONDITIONS: Sjogren's Syndrome
MeSH Terms: conditions — Sjogren's Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sialoscintigraphy (healthy control for nomogram) (Other): Healthy population for nomogram of sialoscintigraphy
  Interventions: Radiation: Sialoscintigraphy
- Sialoscintigraphy (sicca patients) (Other): Patients with sicca symptoms. Data of sialoscintigraphy retrieved from medical records.
  Interventions: Radiation: Sialoscintigraphy

INTERVENTIONS:
Radiation: Sialoscintigraphy — Sialoscintigraphy

SUMMARY:
Sjögren's syndrome is a complex autoimmune disorder. The investigators hypothesize that striated ductal cells may function as non-professional antigen-presenting cells in Sjögren's syndrome. However, there are currently no established methods to assess the functional status of striated ductal cells or their relationship with clinical presentations. To address this knowledge gap, the investigators aim to investigate the potential of sialoscintigraphy, a non-invasive imaging technique, to evaluate the functional status of striated ductal cells. The sodium iodide symporter (NIS), predominantly expressed in striated ductal cells, facilitates the transport of technetium-99m, a radiotracer used in sialoscintigraphy. The investigators hypothesize that the expression level of NIS, as evaluated through sialoscintigraphy, may serve as an indicator of striated ductal cell function and potentially correlate with clinical manifestations in Sjögren's syndrome. However, the literature and our preliminary data lead us to hypothesize that age and the specific major salivary gland being evaluated may introduce confounding factors in the interpretation of sialoscintigraphy results. The investigators therefore proposed to 1) establish a nomogram of sialoscintigraphy stratified by age and specific salivary glands. The investigators will recruit healthy volunteers to receive sialoscintigraphy for the nomogram; 2) associate the expression level of NIS in the striated ductal cells from the major salivary glands with sialoscintigraphy, markers of antigen presentation, and disease manifestations of Sjögren's syndrome. The outcomes will help further applications of sialoscintigraphy in Sjögren's syndrome and formulate hypotheses to explore the pathological mechanisms underlying Sjögren's syndrome.

DETAILED DESCRIPTION:
Sjögren's syndrome is a complex autoimmune disorder characterized by CD4 T lymphocyte infiltration into the salivary glands, leading to impaired glandular function. The mechanisms underlying lymphocyte accumulation and activation in the absence of definitive antigen-presenting cells remain poorly understood. The investigators hypothesize that striated ductal cells, the primary target of lymphocyte invasion, may function as non-professional antigen-presenting cells in Sjögren's syndrome. However, there are currently no established methods to assess the functional status of striated ductal cells or their relationship with clinical presentations. To address this knowledge gap, the investigators aim to investigate the potential of sialoscintigraphy, a non-invasive imaging technique, to evaluate the functional status of striated ductal cells. The sodium iodide symporter (NIS), predominantly expressed in striated ductal cells, facilitates the transport of technetium-99m, a radiotracer used in sialoscintigraphy. The investigators hypothesize that the expression level of NIS, as evaluated through sialoscintigraphy, may serve as an indicator of striated ductal cell function and potentially correlate with clinical manifestations in Sjögren's syndrome. However, the literature and our preliminary data lead us to hypothesize that age and the specific major salivary gland being evaluated may introduce confounding factors in the interpretation of sialoscintigraphy results. Therefore, to address these hypotheses, our research proposal consists of three aims. First, establishing a nomogram of sialoscintigraphy stratified by age and specific salivary glands. The investigators will recruit healthy volunteers to receive sialoscintigraphy for the nomogram. This nomogram will provide a valuable reference for clinical application and further research in interpreting sialoscintigraphy results. Second, associating the expression level of NIS in the striated ductal cells from the major salivary glands with sialoscintigraphy, markers of antigen presentation, and disease manifestations of Sjögren's syndrome. The outcomes will help further applications of sialoscintigraphy in Sjögren's syndrome and formulate hypotheses to explore the pathological mechanisms underlying Sjögren's syndrome. Third, evaluating the capability of antigen presentation in striated ductal cells of salivary glands and to identify potential therapeutic targets. The investigators will examine their ability to uptake extracellular substances and validate their antigen-presenting ability using OT-II cells. Additionally, the investigators will perform RNA sequencing to identify potential therapeutic targets and manipulate their expression to evaluate their impact on the activation of OT-II cells. These findings will confirm that the striated ductal cells as non-professional antigen-presenting cells in Sjögren's syndrome and identify potential therapeutic genetic targets. Overall, our proposed research has the potential to utilize available diagnostic methods to evaluate the striated ductal cells, advance the understanding of how the non-professional antigen-presenting cells participate in the pathogenesis of Sjögren's syndrome, and contribute to the development of innovative therapies.

ELIGIBILITY:
Inclusion Criteria:

* Nomogram: no sicca symptoms
* Sicca: already receiving sialoscintigraphy

Exclusion Criteria (generally):

* pregnancy
* breast feeding
* HIV
* cancer with active treatment

(for nomogram)

* chronic illness needed regular follow-up
* Use anti-histamine, diuretics, anti-depressants, psychotropic medications, anxiolytics or NSAIDs that interfering saliva secretion
* smoking in recent one year
* Positive profiles for anti-SSA or anti-ENA

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Quantitative profiles of sialoscintigraphy, including accumulation velocity and secretion velocity | 3 months within enrollment
  For establishment of sialoscintigraphy nomogram

CONTACTS AND LOCATIONS:
Overall Officials: National Taiwan University Hospital, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No